CLINICAL TRIAL: NCT00239148
Title: A Randomized, Double-blind, Controlled Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Profile and Effects of Repeated Subcutaneous Doses of E1 in Combination With G1 in Type 1 Diabetes
Brief Title: A Study in Type 1 Diabetic Patients With Repeated Doses of E1 in Combination With G1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: INT-201
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — methyl N-acetylsibirosaminide

INTERVENTIONS:
Drug: E1 and G1

SUMMARY:
The purpose of the study is to determine whether E1 and G1 are safe and effective in the treatment of type 1 diabetes.

Type 1 diabetes is an autoimmune disease, in which the immune system attacks pancreatic beta cells. These cells produce insulin, which regulates blood glucose. The mainstay of current treatment for type 1 diabetes is dietary control and daily parenteral administration of insulin.

Recent diabetes research has increasingly focused on pancreatic islet cell replacement, either by islet cell transplantation or by endogenous regeneration of islet cells. During fetal development, islet precursor cells proliferate and differentiate into mature beta cells capable of producing insulin. This process is known as islet cell neogenesis. Islet cell neogenesis normally ceases around birth, however, the adult pancreas still retains significant potential for islet regeneration, as shown by tissue repair following pancreatic injury. Pre-clinical studies have shown that E1 and G1 can re-establish islet cell neogenesis and increase pancreatic insulin production in diabetic animal models. It is therefore postulated that treatment with E1 and G1 may produce islet cell regeneration in type 1 diabetic patients.

DETAILED DESCRIPTION:
In this study, 20 type 1 diabetic patients requiring insulin therapy will be randomized. Fifteen (15) patients will be randomized to receive active study medication and 5 patients will be randomized to receive vehicle control. After undergoing screening procedures, potential patients will enter a 14 day baseline phase where baseline data will be collected. Pending successful completion of the baseline phase, patient will enter a 28-day treatment phase where they will be randomized to receive either once daily subcutaneous injections of E1 plus G1, as separate injections or once daily subcutaneous injections of vehicle control (as 2 separate injections). Patients will receive once daily doses in the morning after breakfast for a period of 28 days. Upon completion of treatment, all patients will continue in the follow-up phase for an additional 6 months and will return to the clinic for monthly visits. Throughout the study, patients will remain on their insulin regimen and will maintain a diary record of insulin intake and blood glucose levels.

Pancreatic beta cell function or insulin secretion is best measured by determination of c-peptide (which is co-secreted with insulin in a 1:1 ratio). An arginine stimulated c-peptide test will therefore be performed at frequent intervals during the study. Patients will be injected with a solution containing arginine, a normal constituent of food that increases insulin release from beta cells into the blood. After the injection seven blood samples for c-peptide tests will be collected over 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis Type 1 diabetes requiring treatment with insulin for a minimum of 1 year
* On a stable insulin regimen for at least 60 days prior to screening
* Currently self monitoring blood glucose levels at least 3 times per day
* No episodes of severe hypoglycemia for 60 days prior to screening
* Body mass index within the range 19-30 kg/m2
* Patient cannot live alone during the treatment phase and up to 1 month in follow-up

Exclusion Criteria:

* Known of suspected history of significant liver, or other GI disease
* History of significant cardiovascular disease including stroke, peripheral vascular disease or any related symptoms
* History of peptic ulcer disease and/or GI bleeding/perforation
* History of cancer
* History or presence of proliferative retinopathy, severe non-proliferative retinopathy, macular edema or presence of untreated diabetic eye disease
* History of treated peripheral or autonomic neuropathy
* Serum creatine superior or equal to 2.0 mg/dL
* History of hypoglycemia unawareness
* Non-healed diabetic ulcer

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of repeated subcutaneous doses of E1 in combination with G1 in patients with type 1 diabetes

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic (PK) profile and clinical effects of repeated subcutaneous doses of E1 in combination with G1 in patients with type 1 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Pastrak, M.D., Study Director — OPKO Health, Inc.
Locations (5):
- United States (5):
  - Pinnacle Research Group, Anniston, Alabama
  - Diablo Clinical Research, Walnut Creek, California
  - Diabetes - Endocrinology Center of West New York, Buffalo, New York
  - Highgate Specialty Center, Durham, North Carolina
  - Diabetes and Glandular Disease Research Associates, San Antonio, Texas